CLINICAL TRIAL: NCT02593656
Title: Effects of Frequent, High Quality, Multi-Ingredient Protein Meals and Exercise Training on Hormones, Body Composition, Muscular Performance, and Energy Metabolism in Active Healthy Men and Women
Brief Title: Effects of Protein Ingestion and Exercise Training on Muscular Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1401-382
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Physical Performance
Keywords: protein ingestion; resistance exercise; interval exercise; stretching exercise; endurance exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Protein (Experimental): Ingestion of 2.0 grams of protein per kilogram of body weight per day combined with exercise training
  Interventions: Behavioral: High Protein
- Normal Protein (Active Comparator): Ingestion of 1.0 gram of protein per kilogram of body weight per day combined with exercise training
  Interventions: Behavioral: Normal Protein

INTERVENTIONS:
Behavioral: High Protein — Protein-pacing throughout the day and exercise training for 12 weeks
  Arms: High Protein
Behavioral: Normal Protein — Normal protein intake throughout the day and exercise training for 12 weeks
  Arms: Normal Protein

SUMMARY:
This study systematically quantified the effects of a protein pacing energy and performance (IEPS) meal pattern compared to a standard recommended control (C) diet both of which were combined with a 4-day/week exercise training program on total and regional (abdominal) body composition (lean mass and fat mass), muscular strength and performance, flexibility, blood lipids and glucose, hormones, mood state and energy metabolism in 60 healthy middle-aged (25-55 years old) men and women following a 12-week intervention. Participants were enrolled in one of two cohorts:

1. Experimental, 2g/kg/Body Weight (BW) Protein (IEPS) (n=30)
2. Control, 1g/kg/Body Weight Protein (C) (n=30)

DETAILED DESCRIPTION:
Participants were matched for body weight, body mass index (BMI) and percent body fat (%BF) and then randomly assigned to one of two groups: (1) Experimental 2.0 g/kg Body Weight per day of protein and combined exercise training (IEPS, n=30); or (2) a control (C) diet containing 1.0 g/kg Body Weight per day of protein and combined exercise training (C, n=30). All participants followed a program of progressive exercise training for 12 weeks performed either in the early morning (0600-0800, AM) or evening (1830-2030, PM). All testing procedures (see below) were administered pre-intervention and post intervention.

Participants in both groups were provided meal plans and instructed to follow the meal plans throughout the intervention. Participants in the IEPS were provided two shakes and 1 bar meal replacement each day to help them meet the 2.0 g/kg Body Weight of protein per day. Participants were given a 2-wk supply of the supplement and asked to return the empty packets before they received the next two-week's supply as a means of assessing their compliance. C participants were required to follow a healthy meal plan providing 1.0 g/kg Body Weight of protein per day by consuming whole foods for all of their meals. They were not provided additional protein supplements. However, they were provided food supplies consisting of granola bars, chocolate milk, and fruit to help them meet their 1.0 g/kg BW protein per day. They were also asked to return empty food packets to monitor compliance. Similar dietary interventions to the two proposed in this study have been used successfully in the past by the PI with no adverse events being reported.

Prior to the start of the study, each subject was familiarized with the exercise training protocols by participating in eight supervised exercise sessions over a two-week period (4 times per week) in the Skidmore College fitness and weight training rooms located adjacent to the Health & Exercise Sciences Department. Participants were asked to perform all the exercise sessions at Skidmore College for the first two weeks and had the option to perform one or two of the exercises (I, E) on their own at home or at their local gym following the two week familiarization. Participants were required to perform 4 exercise sessions per week of the following exercises: a) resistance training (R); b) interval sprint training (I); c) stretching training (S); and d) endurance training (E). During the course of the interventions, a member of the research team periodically "checked-in" (weekly) with each participant by phone, email, or in-person to answer any questions or provide guidance with the exercise and dietary intake. All exercise training guidelines and recommendations followed the American College of Sports Medicine, such that their exercise intensity will be based on their individual fitness level and health status.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be non-smoking, healthy, men and women with no known cardiovascular or metabolic diseases as assessed by a medical history and approval by their physicians to participate. All participants will be active (>30 min, 4d/wk of structured physical activity > 3 years) as assessed by a Physical Activity questionnaire, normal weight (BMI=20-27.5 kg/m2; % body fat<30%), middle aged (25-55 years), and weight stable (+/-2kg) for at least 6 months prior to beginning the study

Exclusion Criteria:

* Individuals will be excluded from participation for the following reasons: orthopedic conditions that preclude or limit participation in the exercise training (RISE); history of cardiometabolic disease (e.g., diabetes, heart disease, etc.) and/or cancer; pregnant or may be pregnant; or allergic to milk products.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Muscular Strength and Power | baseline and post 12 week intervention
  Changes in one repetition muscular strength and power of upper and lower body

SECONDARY OUTCOMES:
Total and Regional Body Composition | baseline and post 12 week intervention
  Changes in total and abdominal body fat and lean body mass by dual energy xray

OTHER OUTCOMES:
Arterial function | baseline and post 12 week intervention
  Changes in arterial stiffness
Blood Lipids | baseline and post 12 week intervention
  Changes in total, LDL, and HDL cholesterol
Energy Metabolism | baseline and post 12 week intervention
  Changes in resting metabolic rate and substrate utilization via indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Arciero, Phd, Principal Investigator — Skidmore College